CLINICAL TRIAL: NCT07232420
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of BL-M24D1 for Injection in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer and Other Solid Tumors
Brief Title: A Study of BL-M24D1 in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M24D1-101
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer; Solid Tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-M24D1 (Experimental): Participants receive BL-M24D1 as intravenous infusion for the first cycle (2 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M24D1

INTERVENTIONS:
Drug: BL-M24D1 — Administration by intravenous infusion for a cycle of 2 weeks.

SUMMARY:
This study is an open, multicenter, non-randomized phase I clinical trial to evaluate the safety, tolerability, pharmacokinetic characteristics, and preliminary efficacy of BL-M24D1 in patients with locally advanced or metastatic non-small cell lung cancer and other solid tumors.

DETAILED DESCRIPTION:
The study consists of two phases: a dose escalation phase (Phase Ia) and a dose expansion phase (Phase Ib).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements;
2. Gender unrestricted;
3. Age: ≥18 years and ≤75 years (Phase Ia); ≥18 years (Phase Ib);
4. Expected survival time ≥3 months;
5. Locally advanced or metastatic non-small cell lung cancer and other solid tumors;
6. Agree to provide archived tumor tissue specimens or fresh tissue samples from primary or metastatic lesions within the past 3 years;
7. Must have at least one measurable lesion meeting the RECIST v1.1 criteria;
8. ECOG performance status score of 0 or 1;
9. Toxicities from prior antitumor therapy have recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. Organ function levels must meet the requirements;
12. Coagulation function: international normalized ratio ≤1.5, and activated partial thromboplastin time ≤1.5 × ULN;
13. Urine protein ≤2+ or ≤1000mg/24h;
14. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before starting treatment, serum pregnancy must be negative, and they must not be breastfeeding; all enrolled patients (regardless of gender) should use adequate barrier contraception throughout the treatment cycle and for 6 months after treatment ends.

Exclusion Criteria:

1. Use of chemotherapy, biotherapy, or immunotherapy within 4 weeks or 5 half-lives prior to the first dose;
2. History of severe heart disease;
3. QT interval prolongation, complete left bundle branch block, or third-degree atrioventricular block;
4. Active autoimmune or inflammatory diseases;
5. Diagnosis of other malignancies within 5 years prior to the first dose;
6. Hypertension poorly controlled by two antihypertensive medications;
7. Poorly controlled blood glucose;
8. Unstable thrombotic events requiring therapeutic intervention within 6 months prior to the first dose;
9. Lung diseases graded ≥3 according to CTCAE v5.0;
10. Symptoms of active central nervous system metastasis;
11. History of allergy to recombinant humanized antibodies or human-mouse chimeric antibodies, or allergy to any excipient of BL-M24D1;
12. Previous organ transplantation or allogeneic hematopoietic stem cell transplantation;
13. Cumulative dose of anthracyclines >360 mg/m² in previous (neo)adjuvant anthracycline therapy;
14. Positive human immunodeficiency virus antibody, active tuberculosis, active hepatitis B virus infection, or active hepatitis C virus infection;
15. History of interstitial lung disease requiring hormonal treatment, or current ILD;
16. Active infection requiring systemic treatment within 4 weeks prior to the first investigational drug dose;
17. Pleural, peritoneal, pelvic, or pericardial effusion requiring drainage and/or accompanied by symptoms within 4 weeks prior to the first investigational drug dose;
18. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks prior to the first investigational drug dose;
19. Participation in another clinical trial within 4 weeks prior to the first dose;
20. Pregnant or lactating women;
21. Other conditions deemed by the investigator as unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 28 days after the first dose
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ia: Maximum tolerated dose (MTD) | Up to 28 days after the first dose
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle.
Phase Ib: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-M24D1.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M24D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M24D1.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-M24D1 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of BL-M24D1 will be investigated.
T1/2 | Up to approximately 24 months
  Half-life (T1/2) of BL-M24D1 will be investigated.
AUC0-t | Up to approximately 24 months
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL (Clearance) | Up to approximately 24 months
  CL in the serum of BL-M24D1 per unit of time will be investigated.
Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of BL-M24D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Frequency of anti-BL-M24D1 antibody (ADA) will be investigated.
Phase Ib: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Phase Ib: Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Phase Ib: Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China